CLINICAL TRIAL: NCT02235935
Title: The Effect of Hyperbaric Chamber Treatment on Patients With Diabetic Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 112/14
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Does Hyperbaric Chaber Treatment Improve Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetic patients, hyperbaric chamber, diabetic retinopathy

SUMMARY:
Diabetic retinopathy (DR) is a common complication of diabetes and is divided into non proliferative DR and proliferative DR. The damage is caused by either macular edema, macular ischemia that can be followed by vascular proliferation.

Hyperbaric chamber treatment assists in increasing the amount of oxygen in the plasma and in the tissues and has been proven to be beneficial in treating different wounds in diabetic patients but its effect hasn't been tested in diabetic retinopathy yet.

This study will recruit 40 diabetic patients who are scheduled for hyperbaric treatment due to different indications such as chronic wounds or radiation damages and who also have diabetic retinopathy. These patients will undergo opthalmic physical examination including fundus photography and OCT (Optical Coherence Tomography - optical IR retinal photography). Screening for these patients will be conducted at the Hyperbaric chamber at Assaf Harofe Medical Center for all diabetic patients prior to their first treatment.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

1. Patients between ages 18-90 with Diabetes type I or II and diabetic retinopathy who are scheduled for hyperbaric treatment for other indications than DR.
2. Patients who signed an informed consent form and agree to undergo an ophthalmic physical examination, Fundus photography and OCT prior to hyperbaric treatment and oCT exam following every 10 treatments in hyperbaric chamber. Total number of hyperbaric treatments will be conducted according to the main indication for which they have been assigned this treatment.

Exclusion Criteria:

1. Patients with Carotid stenosis of more than 70%
2. Anemia of < 10mg/Dl
3. Patients with chest X ray pathology which cannot be admitted to hyperbaric chamber treatment.
4. Patients with claustrophobia or that cannot decompress properly.
5. Patients with any malignant disease
6. Patients with inability to sign informed consent

Decompression treatment will last 90 minutes in 2 atmospheres pressure with 100% oxygen.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any diabetic patient undergoing hyperbaric chamber treatment due to diabetic ulcers
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
OCT results | 1 month
  the reduction in retina width as recorded on OCT following 20 treatments in Hyperbaric Chamber

SECONDARY OUTCOMES:
Visual Acuity | 1 month
  changes in visual acuity as recorded in ophthalmologic exam before and after treatments in hyperbaric chamber

CONTACTS AND LOCATIONS:
Overall Officials: Shai Efrati, Principal Investigator — Assaf Harofe MC
Locations (1):
- Assaf Harofe Medical Center, Ẕerifin, Israel